CLINICAL TRIAL: NCT01059981
Title: Analysis of Emergency Department Volumes During Natural Disasters
Brief Title: Analysis of Emergency Department (ED) Volumes During Natural Disasters
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: James McCarthy, MD, University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-08-0656
Record Dates: First submitted 2009-02-04; First posted 2010-02-01 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Dialysis; Trauma Related Injuries; Carbon Monoxide Poisoning
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Dialysis patients
- 2: Trauma patients
- 3: Patients with carbon monoxide poisoning

SUMMARY:
The 'Analysis of Emergency Department Volumes during Natural Disasters' retrospective study focuses on three specified populations including dialysis patients, trauma patients, and patients poisoned by carbon monoxide. These three populations have one commonality - hurricanes, ie. natural disasters, which is the exposure. Causal associations and significant correlations will be explored in all three subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carbon monoxide poisoning in addition to trauma and dialysis patients admitted to the Memorial Hermann Health System's (MHHS) Emergency Department (ED) 1 week pre- and post-Hurricane Ike's landfall to the City of Houston, which was September 12, 2008.

Exclusion Criteria:

* Patients with the specified conditions that were not admitted during the time interval allotted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Three populations: Dialsysis patients, trauma patients, and patients experiencing carbon monoxide poisonings during natural disasters.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J McCarthy, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Memorial Hermann Hospital - Medical Center, Houston, Texas
  - University of TX Health Science Center, Houston, Houston, Texas